CLINICAL TRIAL: NCT05964192
Title: Added Value of a Neuroendocrine Test Battery in the Response to Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment : a Pilot Study in Major Depression (Endo-rTMS)
Brief Title: Added Value of a Neuroendocrine Test Battery in the Response to Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment
Acronym: Endo-rTMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Rouffach (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A00288-37
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2023-07

CONDITIONS: Major Depression
Keywords: Depression; clinical outcome; rTMS (repetitive transcranial magnetic stimulation); theta burst; TRH (thyreoliberin) test; DST (dexamethasone suppression test)
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment resistant major depressed inpatients (TRDs) (Experimental)
  Interventions: Procedure: Repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Procedure: Repetitive transcranial magnetic stimulation (rTMS) — The theta burst stimulation (TBS) technique consists in administering bursts of transcranial magnetic stimulation (TMS) at very high frequency (50Hz) for 5 minutes (3 pulses of stimulation given at 50 hz; 10 bursts/1 s train; inter-train interval : 8 s; number of trains : 30; 100% resting motor threshold; number pulses/session : 900). Total number of sessions : 20 sessions (single daily session).

SUMMARY:
The primary objective of the study is to determine the predictive value of the neuroendocrine tests TRH-∆∆TSH (thyreoliberin - thyreostimulin) and DST (dexamethasone suppression test) in the subsequent response to rTMS-TBS (repetitive transcranial magnetic stimulation-theta burst stimulation) treatment, defined as at least a 50% decrease in depression score after 20 sessions of rTMS-TBS.

DETAILED DESCRIPTION:
Conduct of research :

This is a monocentric, non-randomized, open-label pilot study involving 50 male and female patients aged 18 to 65, hospitalized for major depression and presenting with an indication for treatment with repeated theta-burst transcranial magnetic stimulation (rTMS-TBS), i.e. a situation of therapeutic failure following 2 well-conducted antidepressant treatments.

At the end of the 20 rTMS-TBS sessions (one session per day, except weekends), the clinical response will be assessed by an investigator "blind" to the endocrine results. This response will be analyzed according to the status of neuroendocrine tests at inclusion (TRH-∆∆TSH and DST) and at the end of the study (for those who had one or more abnormal tests at inclusion and in whom the same tests were repeated at the end of the rTMS-TBS sessions).

During the inclusion visit, the patient and investigator sign the consent form, after double-checking the inclusion and non-inclusion criteria.

Immediately after the tenth rTMS session, an assessment of depression using the HAMD (17-item Hamilton Depression Scale) scale will be carried out by an independent psychiatrist, blind to the results of the neuroendocrine tests. This psychiatrist, who has already administered the HAMD at V0, will repeat the assessments at V1 and V2.

Immediately after the twentieth rTMS session, an assessment of depression using the HAMD scale will be carried out by an independent psychiatrist. This assessment will determine responder/non-responder status to rTMS-TBS.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a characterized depressive episode defined according to DSM-5 (diagnostic and statistical manual of mental disorders) criteria;
2. Patient between the ages of 18 and 65 years;
3. Inpatient with an inadequate response to two prior well-conducted antidepressant treatments (Hamilton 17-item scale [HAMD-17] score at inclusion≥ 18) ;
4. Patient with written informed consent to participate in the study;
5. Patient enrolled in or receiving social security benefits.

Exclusion Criteria:

1. Patient with endocrinopathy ;
2. Patient with a contraindication to neuroendocrine testing (hypersensitivity to the active substance or to one of the excipients);
3. Patient with a contraindication to rTMS:

   * cochlear implant,
   * cardiac pacemaker,
   * metal clips, stents or other electronic implants within one meter of the stimulation coil,
   * intracranial hypertension,
   * poorly balanced comitiality,
   * in the case of well-balanced comitiality, a neurological consultation with electroencephalogram (EEG) is planned before including the patient;
4. Patient previously treated with monoamine oxidase inhibitor (MAOI) antidepressant or lithium salts (within 6 months prior to inclusion);
5. Pregnant or lactating patient;
6. Patient under court protection or deprived of liberty;
7. Patient under guardianship/guardianship.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
17-item Hamilton Depression Scale (HAMD) | Change from inclusion result at 6 weeks (after 20 rTMS-TBS sessions)
  Clinical response will be defined by at least a 50% decrease in depression score at the end of the 20 rTMS-TBS sessions - measured by the 17-item Hamilton Depression Scale (HAMD) - compared to inclusion (Carrozzino et al, 2020). The predictive value of the TRH-∆∆TSH on the one hand, and the DST on the other, will be assessed using an ROC curve and its AUC (Area Under the Curve) calculation.

SECONDARY OUTCOMES:
Hamilton Depression Scale (HAMD) | Through study completion, an average of 6 weeks
  Functional remission will be defined by a HAMD score ≤ 8 at the end of 20 sessions of rTMS-TBS
Evolution of neuroendocrine parameters | Through study completion, an average of 6 weeks
  Pre- and post-treatment difference in neuroendocrine test values
Evolution of neuroendocrine parameters | Through study completion, an average of 6 weeks
  Proportion of patients having normalized their tests at the end of the 20 sessions of rTMs.
Relationship of the therapeutic response with the evolution of neuroendocrine parameters | Through study completion, an average of 6 weeks
  Proportion of responders/functional remission patients according to the normalization or not of neuroendocrine tests after rTMS-TBS treatment.
Predictive factors | Through study completion, an average of 6 weeks
  Predictors of response to rTMS treatment (e.g., demographics)

CONTACTS AND LOCATIONS:
Overall Officials: MIHAELA TOMSA, PhD, Principal Investigator — CENTRE HOSPITALIER DE ROUFFACH
Locations (1):
- Centre Hospitalier Rouffach, Rouffach, Alsace, France

IPD SHARING:
Plan to Share IPD: No